CLINICAL TRIAL: NCT03359525
Title: Prospective Randomized Study Comparing Topical Versus Intravenous Tranexamic Acid in Anterior Total Hip Arthroplasty
Brief Title: Study Comparing Topical Versus Intravenous Tranexamic Acid in Anterior Total Hip Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Samik Banerjee, Principal Investigator, Division of Orthopaedic Surgery, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4744
Record Dates: First submitted 2017-11-15; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Tranexamic Acid Adverse Reaction
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Group A: Intravenous Tranexamic acid at a dose of 1 gram administered 30 min prior to skin incision and 1 gram 3 hours after the procedure. (Total dose administered is 2 grams)
  Interventions: Drug: Tranexamic Acid
- Group B (Experimental): Group B: Topical Tranexamic acid at a dose of 1 gram injected in to the periarticular tissues prior to closure and 1 gram injected into the joint through the drain following wound closure. (Total dose administered is 2 grams)
  Interventions: Drug: Tranexamic Acid
- Group C (Experimental): Group C: Combined Intravenous 1 gram given intravenous 30 min prior to skin incision and topical tranexamic acid (1 gram) injected in to the periarticular tissues prior to closure. (Total dose administered is 2 grams)
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — intravenous versus Intraarticular versus intravenous

SUMMARY:
Brief Summary Title: Prospective Randomized Trial Comparing Topical Versus Intravenous Tranexamic Acid (TXA) in Anterior (Total hip arthroplasty) Several strategies have been used to reduce transfusion requirements during total hip arthroplasty (THA). Recently, anti-fibrinolytic agent TXA, has been used extensively in THAs to minimize intra-operative blood losses. However, few studies have compared the efficacy of topical versus intravenous use in direct anterior THA. Therefore, the investigators will attempt to evaluate differences in the post-operative outcomes of topical versus intravenous TXA in Direct anterior approach to THA. The investigators propose to conduct a prospective randomized study in which patients who have exhausted non-operative treatment for hip osteoarthritis and are opting for THA will be randomized into 3 groups in a 1:1:1 ratio based on a computer generated algorithm following inclusion and exclusion criteria as described below. Patients will be distributed in to 3 groups as follows: Group A: Intravenous TXA at a dose of 1 gram administered 30 min prior to skin incision and 1 gram 3 hours after the procedure. (Total dose: 2 grams) Group B: Topical TXA at a dose of 1 gram injected in to the peri-articular tissues prior to closure and 1 gram injected into the joint through the drain following wound closure. (Total dose:2 grams) Group C: Combined Intravenous 1 gram given intravenous 30 min prior to skin incision and topical TXA (1 gram) injected into the peri-articular tissues prior to closure. (Total dose: 2 grams). The number of subjects needed to achieve 90% power was calculated based on a one-way fixed effects analysis of variance with 3 levels. Primary endpoint used was drainage measured in milliliters in the post-operative (POD) #1 following surgery. Criterion for significance (alpha) was set at 0.05 and the ANOVA statistics was non-directional (two tailed). Preliminary data indicated that drainage volume averages 250 ml with a standard deviation of 160 ml in our operating room. Difference (maximum to minimum of the three levels) of 150 ml was judged to be the minimally clinically relevant difference in drainage volume (effect size =0.38). A 20% loss to follow up was also assumed. The study will need 38 cases per cell for a total of 114 cases to achieve 90% power of detecting a difference this large. Data metrics will be tabulated into excel spreadsheets. Data analysis will be performed using statistical software. Quantitative data will be analyzed using non-directional analysis of variance (ANOVA) with Tukey's test for multiple comparisons. Non-normality or heteroscedasticity of data will either be corrected by transformation or a non-parametric (Kruskal Wallis) test will be used. Categorical data will be analyzed using chi-square tests (or Fisher's exact test if any cells expected value is 5 or less). A p-value <0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
Detailed Description Prospective Randomized Study Comparing Topical versus Intravenous Tranexamic Acid in Anterior Total Hip Arthroplasty A. Study Background and Purpose Hip and knee arthroplasty is one of the most successful procedures for relieving pain and correction of deformity in patients with degenerative arthritis of the hip and knee with approximately 1 million procedures performed every year in the United States. However, these joint replacements are associated with substantial amounts of blood loss varying between 500 and 1,500 milliliters often necessitating allogeneic blood transfusions in the post-operative period. This potentially leads to delays in discharge, physical recovery, and increased complications. In addition, it can escalate the cost of total joint arthroplasties in healthcare organizations. Several strategies have been employed in the past with varying efficacies to reduce transfusion requirements including preoperative autologous donation, erythropoietin use, intra-operative hypotensive anesthesia, fibrin spray, cell salvage, and post-operative auto-transfusions drains. Over the past decade the anti-fibrinolytic agent tranexamic acid, a synthetic analog of the amino acid lysine, has been used extensively in lower extremity arthroplasties to minimize intra-operative blood losses. Tranexamic acid prevents the conversion of plasminogen to plasmin on the surface of fibrin, thereby inhibiting fibrinolysis and reducing blood loss. Despite its almost universal use and documented safety, there is significant controversy regarding the optimal route of administration with several studies documenting equivalent efficacy of intravenous and topical administration, with both routes of administration currently considered standard of care in both hip and knee arthroplasties. Anecdotally, the senior author has found that topical use of tranexamic acid has led to greater post-operative drainage and reduction in hematocrit compared to intravenous use. This may be secondary to the absence of tamponade effect with anterior total hip arthroplasty. However, few studies have compared the efficacy of topical versus intravenous use of this medication in direct anterior total hip arthroplasty. Therefore, in this prospective randomized study, the investigators will attempt to evaluate if there exists any significant difference in the post-operative outcomes of topical versus intravenous tranexamic acid following anterior total hip arthroplasty.

B. Study Design This will be a prospective randomized study in which subjects who have exhausted non-operative treatment for hip osteoarthritis and are opting for total hip arthroplasty will be randomized into 3 groups in a 1:1:1 ratio based on a computer generated algorithm following inclusion and exclusion criteria as described below. The patients will be recruited into the study by the principal investigator from his practice cohort. They will be consented to enroll in to the study by any one of the co-investigators. They will either be recruited in the office at Bone and Joint Center, 1367 Washington Avenue, Albany New York or at Albany Medical Center, 43 New Scotland Avenue on the day of surgery. Patients will be further stratified according to BMI (body mass index) as this may be a confounding variable affecting blood loss. The patients will be distributed in to 3 groups as follows: Group A: Intravenous Tranexamic acid at a dose of 1 gram administered 30 min prior to skin incision and 1 gram 3 hours after the procedure. (Total dose administered is 2 grams); Group B: Topical Tranexamic acid at a dose of 1 gram injected in to the peri-articular tissues prior to closure and 1 gram injected into the joint through the drain following wound closure. (Total dose administered is 2 grams); Group C: Combined Intravenous 1 gram given intravenous 30 min prior to skin incision and topical tranexamic acid (1 gram) injected in to the peri-articular tissues prior to closure. (Total dose administered is 2 grams). Women who are premenopausal will have a pregnancy test prior to total hip arthroplasty as per institutional protocol. This will be covered by the patient's health insurance. Subjects will be assigned a unique identification number. The principal investigators will maintain a list identifying all subjects by their subject identification number and initials. Subjects will be screened at the time of scheduling surgery in the outpatient clinic. Study procedures and information regarding the nature of the study will be reviewed with potential subjects, and written informed consent will be obtained prior to any study-related procedures. Alternatively, patients may be contacted by phone regarding the study. In this case, the study information will be reviewed with the subject over the phone and subjects will be asked to electronically sign a consent form sent via e-mail. Patients will be given a flyer when they are booked for surgery which will briefly outline our study and inform them that they may be contact about the study via telephone. The phone consent will be performed by one of the primary or co-investigators listed on this study. Adobe E-sign software will be used to send subjects a consent form via e-mail after the phone conversation. The patient will be given an opportunity to review the consent document and then the investigator will place a second call to the subject to review any questions or concerns. The subject and the investigator will the electronically sign the consent in succession. The Adobe E-signature software provides a date and time stamp. After the consent is signed by both parties the subject will be provided a copy of the signed consent by email. A copy of the consent will be maintained in a secure network drive provided by Albany Medical Center which will be accessible by the investigators listed on the study. A printed copy of the signed consent will be placed into the patients chart on the date of surgery. A second printed copy will be placed in a locked file cabinet in the preoperative unit at Albany Medical Center. All patients will have the right to voluntarily withdraw from the study. Any intra-operative or post-operative adverse events prior to discharge from the hospital will be recorded.

Other screening procedures are as follows:

i. Review inclusion and exclusion criteria. ii. Collect demographic information including age, sex, weight, height, BMI, American Society of Anesthesiology status, co-morbidities, and medication use.

iii. Record medical history. iv. Collect baseline data with regards to pre-operative hematocrit, creatinine levels, and coagulation profile.

All patients will have combined spinal with 0.75% bupivacaine heavy with lumbar and sacral plexus blocks. The total hip arthroplasties will be performed through a direct anterior approach. A closed suction drain will be placed intra-operatively and daily outputs measured will be recorded. The drain will be clamped in all patients for 1 hour in the immediate post-operative period after wound closure. For group B, the drain will be clamped after 1 gram tranexamic acid is injected through the drain following completion of wound closure. Blood transfusion postoperatively will be dictated by the institutional policy of post-operative hemoglobin concentration of <7 g/dl or hematocrit of <21 or when patients developed any anemia-related organ dysfunction such as alteration of mental status, respiratory distress, or palpitations. The total blood loss will be calculated using a modification of the Gross formula where, if a reinfusion or an allogeneic transfusion was performed, the total blood loss will be equal to the loss calculated from the change in the hematocrit plus the volume transfused 20-22.

Prophylaxis against venous thromboembolism will be administered according to standard practice at our center which includes anti-embolic stockings, intermittent pneumatic compression, and early physical therapy on the day after surgery, aspirin 325 milligrams twice daily started on first post-operative day and continued at discharge. Analgesic irrigation with 7.5 ml of 1% Ropivacaine, 0.25 ml of Epinephrine 1mg/1ml, 1 ml of Morphine 10mg/ml, 1 ml of Ketorolac 30mg/ml, 1 ml of methylprednisolone acetate 40mg/ml, and 60 ml of normal saline will be administered for wound infiltration in the peri-capsular tissues prior to closure unless the patient possesses allergies to any of the aforementioned medications. Post-operatively, all patients (Groups, A, B, and C) will receive standard post-operative analgesic medications. All patients will be discharged with pregabalin 75 mg twice daily (BID), celecoxib 200 mg BID, Oxycodone/acetaminophen 5/325 mg to take 1-2 tabs every four hours as needed for pain control, and aspirin 325 mg BID for thromboprophylaxis unless they possess allergies to the aforementioned medications.

Duration of the study The proposed data collection period of this study is two years. Patients will not be brought back for follow-up beyond their normal post-operative visit schedule. They will be seen earlier if any complications arise. During their visits metrics that will be specifically assessed include wound infections rates and incidences of deep vein thrombosis/ pulmonary thromboembolism (DVT/PE). Emergency department visits and readmissions, if any, will be recorded.

Withdrawal

Any of the subjects may withdraw from the study at any time without prejudice. However, every attempt should be made to encourage subjects to complete the study. If a subject discontinues from the study, the reason given must be fully evaluated and recorded appropriately in source documentation and the electronic health record. If the subject is withdrawn because of an adverse event (AE), that AE must be indicated as the reason for withdrawal. The investigator can discontinue a subject at any time if medically necessary. The primary investigator may replace subjects that are withdrawn. In addition, subjects meeting the following criteria must be withdrawn from the study:

* Occurrence of any adverse event (AE), post-operative bleeding complications requiring return to operating room or a vascular intervention radiology procedure, or laboratory abnormality which, in the opinion of the primary investigator, warrants the subject's permanent withdrawal from the study;
* Subject noncompliance, defined as refusal or inability to adhere to the study schedule;
* At the request of the subject, primary investigator, or regulatory authority
* Subject is lost to follow-up.

C. Subject Population The subjects will be male and female patients of the principal orthopedic surgeon's practice who are eligible for unilateral anterior total hip arthroplasty. They must meet the above stated inclusion criteria and be willing to participate in the study and receive any of the three routes of tranexamic acid. They will be preoperatively evaluated for medical clearance by either their primary care physician and/or cardiologist as they otherwise would regardless of study inclusion.

D. Study Location The study will be conducted at Albany Medical Center, 43 New Scotland Avenue, Albany New York, Zip 12208, (Phone: 518-262-4000) and Bone and Joint Center, 1367 Washington Avenue, Albany New York, 12206 (Phone 518-489-2666).

E. Data analysis All data metrics including demographic variables and primary and secondary endpoints will be tabulated in to an excel spreadsheet (Microsoft Inc., Redmond, WA). Data analysis will be performed using software GraphPad Prism (GraphPad Software Inc., CA). Quantitative data will be analyzed using non-directional analysis of variance (ANOVA) with Tukey's test for multiple comparisons. Non-normality or heteroscedasticity of data will either be corrected by transformation or a non-parametric (Kruskal Wallis) test will be used. Data will be presented as mean and standard deviation if normal or median and interquartile range if not. Categorical data will be analyzed using chi-square tests (or Fisher's exact test if any cells expected value is 5 or less). A p-value <0.05 will be considered statistically significant. Risks of total hip arthroplasty, equally applicable to all participants in the study, include intra-operative fracture, post-operative infection, deep-vein thrombosis, pulmonary embolism, post-operative hip pain, and need for future surgery. Complications associated with the use of tranexamic acid include unforeseen allergic complications.

G. Benefits The primary advantage, which study subjects may derive from being a part of this study include considerable improvements in blood loss in the immediate peri-operative period. The benefit expected for study subjects enrolled in this study may include a reduction in length of stay, fewer blood transfusions, and earlier achievement of rehabilitative outcomes.

H. Confidentiality All primary data, or copies thereof (e.g., laboratory records, data sheets, correspondence, photographs, and computer records), which are a result of the original observations and activities of the study and are necessary for the reconstruction and evaluation of any study report, will be retained by the Principal Investigator. Data sources will be Albany Medical Center Sorian electronic health record and from Electronic health records (EHR) at Bone and Joint Center. The results from screening and data collected during the study will be recorded in the electronic health records and/or source documents, as appropriate, for each subject. To maintain confidentiality, the subjects will be identified by numbers and/or initials on the electronic health records. Beginning on the day of surgery, all patients included in the study will be given a number associated with a randomly assigned opaque envelope. The only association between patients and their assigned numbers will be stored in the principal investigator's locked file cabinet in the locked office. However, as an inpatient, all data will be stored under the patient's name in the medical record in standard fashion. After discharge, data will be copied onto a file by one of the co-investigators and stored under the patient's confidential number. From this point on, all data identifying information will be de-identified from the patient.

I. Options Since intraoperative tranexamic acid use has been shown to be standard of care, option of not using tranexamic acid increases the risks of bleeding and post-operative blood transfusions.

ELIGIBILITY:
Inclusion Criteria

To be eligible to participate in the study, subjects must meet the following criteria:

1. Males or females age > 18 years and <80 years
2. Informed consent
3. Diagnosis of primary osteoarthritis or osteonecrosis
4. Previous history of contralateral hip or knee arthroplasty will not be excluded from the study Exclusion criteria

Subjects who meet any of the following criteria will NOT be eligible to participate in the study:

1. Unable to comply with study requirements i.e unable to complete first follow-up visit at 4 weeks or if they are unable to follow-up.
2. Has an active joint infection\
3. Immuno-suppression, e.g., human immunodeficiency virus (HIV) infection, s/p organ transplantation, receipt of steroids for > 10 days at > 10 mg of prednisone equivalent daily within the 90 days prior to enrollment
4. Chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
5. Body mass index > 45
6. Life expectancy < 6 months
7. Renal insufficiency (serum creatinine >2.5 mg/dl)
8. Pre-operative Hemoglobin <8 gm/dl
9. Congenital and acquired coagulopathy
10. Patients on pre-operative therapeutic anticoagulation
11. Patients who need post-operative therapeutic anticoagulation
12. Pregnancy and nursing mothers or women who are expected to nurse their babies within one month of surgery
13. History of thromboembolism, stroke, transient ischemic attack, traumatic brain injury, subdural, or subarachnoid hemorrhage
14. History of reported allergy to tranexamic acid
15. Uncontrolled Hypertension
16. Non-steroidal antiinflammatory use within 3 weeks of surgery other than Celebrex.
17. Patients who continue the use of aspirin and have not stopped for more than 7 days prior to surgery.
18. Patients who need to be on any anticoagulation other than aspirin 325 mg BID will be excluded from the study.
19. Prisoners will be excluded from the study.
20. Patients with history of acquired defective color vision
21. Plan for staged bilateral total hip procedures within 14 days
22. Family history of thromboembolism
23. Patient unable to receive spinal anesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative drain output | Drain output will be measured in milliliters on Post-operative Day 1 following total hip arthroplasty . This will be a one time measurement for every participant enrolled in the study.
  This will be measured from the drain output recorded over 24 hours on Post-operative day 1. This is a one time measurement for every participant enrolled in to the study.

SECONDARY OUTCOMES:
Change in post operative hemoglobin | Post-operative day 1 and day 2 hemoglobin change compared to pre-operative hemoglobin.
  calculated from change in pre-op and post operative hemoglobin measured in g/dl. There will be 2 recordings for every participant enrolled in the study for the entire study period.
Allogeneic blood transfusion rates | Measured in the number of participants had transfusion during first week following total hip arthroplasty
  Measured in the number of participants who received a blood transfusion during the hospital stay following total hip arthroplasty
Readmissions | Number of readmissions and emergency department visits measured in number of patients who were readmitted or visited the emergency department during first 90 days after surgery.
  Number of times participants were admitted after the surgery within 90 days after surgery
Length of stay | Measured in number of days patient stayed in the hospital following total hip arthroplasty. This will be one measurement for each participant in the study within 1 week after surgery.
  Number of days the patient spent in the hospital after total hip arthroplasty
DVT | Incidence of deep vein thrombosis measured in number of patients having this complication during first 90 days after surgery
  Incidence of DVT among participants enrolled in the study occurring with 90 days of surgery.
Wound infection | Wound infection rates measured in number of cases occuring within first 90 days after total hip arthroplasty.
  Incidence of superficial and deep wound infection among participants enrolled in the study
Emergency department visits | Number of times participants visited the emergency department after discharge from the hospital within 90 days after total hip arthroplasty
  Number of times participants visited the emergency department after discharge from the hospital within 90 days after total hip arthroplasty
Pulmonary Thromboembolism | Incidence of Pulmonary thromboembolism measured in number of patients having this complication during first 90 days after surgery
  Incidence of Pulmonary thromboembolism among participants enrolled in the study occurring with 90 days of surgery.
Number of units of blood transfused | Measured in the number of units of blood transfusion the participants received during the first week following total hip arthroplasty.
  Measured in the number of units of blood transfusion each participant received a blood transfusion during their hospital stay following total hip arthroplasty.
Change in post operative hematocrit compared to pre-operative hematocrit | Post-operative day 1 and day 2 hematocrit change compared to pre-operative hematocrit.
  calculated from change in pre-op and post op hematocrit measured in percentage. There will be 2 recordings for every participant enrolled in the study for the entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: Ravneet S Bhullar, MD, Principal Investigator — Albany Medcial Center
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Result] Carling MS, Jeppsson A, Eriksson BI, Brisby H. Transfusions and blood loss in total hip and knee arthroplasty: a prospective observational study. J Orthop Surg Res. 2015 Mar 28;10:48. doi: 10.1186/s13018-015-0188-6. PMID 25889413
- [Result] Kasparek MF, Faschingbauer M, Waldstein W, Boettner CS, Boettner F. Topical Tranexamic Acid is Equivalent to Targeted Preoperative Autologous Blood Donation in Total Hip Arthroplasty. J Arthroplasty. 2017 Apr;32(4):1176-1179. doi: 10.1016/j.arth.2016.10.026. Epub 2016 Oct 31. PMID 27913130
- [Result] Shang J, Wang H, Zheng B, Rui M, Wang Y. Combined intravenous and topical tranexamic acid versus intravenous use alone in primary total knee and hip arthroplasty: A meta-analysis of randomized controlled trials. Int J Surg. 2016 Dec;36(Pt A):324-329. doi: 10.1016/j.ijsu.2016.11.033. Epub 2016 Nov 14. PMID 27856355
- [Result] Moskal JT, Capps SG. Meta-analysis of Intravenous Tranexamic Acid in Primary Total Hip Arthroplasty. Orthopedics. 2016 Sep 1;39(5):e883-92. doi: 10.3928/01477447-20160526-02. Epub 2016 Jun 1. PMID 27248332
- [Result] Anand A, Melvin JS. Tranexamic Acid in Hip and Knee Arthroplasty. J Am Acad Orthop Surg. 2016 Jun;24(6):e59. doi: 10.5435/JAAOS-D-15-00708. No abstract available. PMID 27135795
- [Result] Wei Z, Liu M. The effectiveness and safety of tranexamic acid in total hip or knee arthroplasty: a meta-analysis of 2720 cases. Transfus Med. 2015 Jun;25(3):151-62. doi: 10.1111/tme.12212. Epub 2015 May 29. PMID 26033447
- [Result] Wang C, Xu GJ, Han Z, Ma JX, Ma XL, Jiang X, Wang Y. Topical application of tranexamic acid in primary total hip arthroplasty: a systemic review and meta-analysis. Int J Surg. 2015 Mar;15:134-9. doi: 10.1016/j.ijsu.2014.12.023. Epub 2015 Jan 7. PMID 25576011
- [Result] Wu YG, Zeng Y, Yang TM, Si HB, Cao F, Shen B. The Efficacy and Safety of Combination of Intravenous and Topical Tranexamic Acid in Revision Hip Arthroplasty: A Randomized, Controlled Trial. J Arthroplasty. 2016 Nov;31(11):2548-2553. doi: 10.1016/j.arth.2016.03.059. Epub 2016 Apr 12. PMID 27179770
- [Result] Poeran J, Rasul R, Suzuki S, Danninger T, Mazumdar M, Opperer M, Boettner F, Memtsoudis SG. Tranexamic acid use and postoperative outcomes in patients undergoing total hip or knee arthroplasty in the United States: retrospective analysis of effectiveness and safety. BMJ. 2014 Aug 12;349:g4829. doi: 10.1136/bmj.g4829. PMID 25116268
- [Result] Madsen RV, Nielsen CS, Kallemose T, Husted H, Troelsen A. Low Risk of Thromboembolic Events After Routine Administration of Tranexamic Acid in Hip and Knee Arthroplasty. J Arthroplasty. 2017 Apr;32(4):1298-1303. doi: 10.1016/j.arth.2016.10.015. Epub 2016 Oct 20. PMID 27843042
- [Result] Hanna SA, Prasad A, Lee J, Achan P. Topical Versus Intravenous Administration of Tranexamic Acid in Primary Total Hip Arthroplasty: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Orthop Rev (Pavia). 2016 Sep 19;8(3):6792. doi: 10.4081/or.2016.6792. eCollection 2016 Sep 19. PMID 27761223
- [Result] Chen Y, Chen Z, Cui S, Li Z, Yuan Z. Topical versus systemic tranexamic acid after total knee and hip arthroplasty: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2016 Oct;95(41):e4656. doi: 10.1097/MD.0000000000004656. PMID 27741100
- [Result] Hallstrom B, Singal B, Cowen ME, Roberts KC, Hughes RE. The Michigan Experience with Safety and Effectiveness of Tranexamic Acid Use in Hip and Knee Arthroplasty. J Bone Joint Surg Am. 2016 Oct 5;98(19):1646-1655. doi: 10.2106/JBJS.15.01010. PMID 27707851
- [Result] Li J, Zhang Z, Chen J. Comparison of efficacy and safety of topical versus intravenous tranexamic acid in total hip arthroplasty: A meta-analysis. Medicine (Baltimore). 2016 Sep;95(36):e4689. doi: 10.1097/MD.0000000000004689. PMID 27603364
- [Result] Babis GC. Controversy in Tranexamic Acid Administration Route Continues: Commentary on an article by Zeng Yi, MD, et al.: "Tranexamic Acid Administration in Primary Total Hip Arthroplasty: A Randomized Controlled Trial of Intravenous Combined with Topical Versus Single-Dose Intravenous Administration". J Bone Joint Surg Am. 2016 Jun 15;98(12):e51. doi: 10.2106/JBJS.16.00128. No abstract available. PMID 27307369
- [Result] Yi Z, Bin S, Jing Y, Zongke Z, Pengde K, Fuxing P. Tranexamic Acid Administration in Primary Total Hip Arthroplasty: A Randomized Controlled Trial of Intravenous Combined with Topical Versus Single-Dose Intravenous Administration. J Bone Joint Surg Am. 2016 Jun 15;98(12):983-91. doi: 10.2106/JBJS.15.00638. PMID 27307358
- [Result] Kang JS, Moon KH, Kim BS, Yang SJ. Topical administration of tranexamic acid in hip arthroplasty. Int Orthop. 2017 Feb;41(2):259-263. doi: 10.1007/s00264-016-3195-2. Epub 2016 Apr 18. PMID 27087627
- [Result] North WT, Mehran N, Davis JJ, Silverton CD, Weir RM, Laker MW. Topical vs Intravenous Tranexamic Acid in Primary Total Hip Arthroplasty: A Double-Blind, Randomized Controlled Trial. J Arthroplasty. 2016 Apr;31(4):928-9. doi: 10.1016/j.arth.2015.12.001. Epub 2015 Dec 17. No abstract available. PMID 26783121
- [Result] North WT, Mehran N, Davis JJ, Silverton CD, Weir RM, Laker MW. Topical vs Intravenous Tranexamic Acid in Primary Total Hip Arthroplasty: A Double-Blind, Randomized Controlled Trial. J Arthroplasty. 2016 May;31(5):1022-6. doi: 10.1016/j.arth.2015.11.003. Epub 2015 Nov 10. PMID 26703193
- [Result] Gross JB. Estimating allowable blood loss: corrected for dilution. Anesthesiology. 1983 Mar;58(3):277-80. doi: 10.1097/00000542-198303000-00016. No abstract available. PMID 6829965
- [Result] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146
- [Result] Liu X, Zhang X, Chen Y, Wang Q, Jiang Y, Zeng B. Hidden blood loss after total hip arthroplasty. J Arthroplasty. 2011 Oct;26(7):1100-5.e1. doi: 10.1016/j.arth.2010.11.013. Epub 2011 Jan 21. PMID 21256705